CLINICAL TRIAL: NCT06173752
Title: Leveraging Machine Learning Approaches to Understand Mechanisms of Exposure Therapy in Real-World Settings
Brief Title: Mechanisms of Exposure Therapy for OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Jennie M. Kuckertz, PhD, Research Psychologist, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P003369
Record Dates: First submitted 2023-12-06; First posted 2023-12-18 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exposure therapy (Experimental): Participants will complete exposure therapy for up to 12 weeks, and each coached exposure session will be approximately 50 minutes. Exposure plans will be developed collaboratively between participants and their clinician at the beginning of treatment, and refined iteratively as clinically appropriate. In each coached exposure, participants will:
  1. Complete an Exposure Feedback Form
  2. Wear a wristwatch that provides psychophysiological data
  The intervention will occur across two study sites (McLean Hospital, San Diego State University). Sites will differ on level of care. At McLean Hospital, participants will be recruited from the OCD Institute and will receive exposure therapy via partial hospital or residential setting as part of their standard care, regardless of participation in the study. At San Diego State University, participants will be recruited to receive exposure therapy via outpatient setting.
  Interventions: Behavioral: Exposure therapy

INTERVENTIONS:
Behavioral: Exposure therapy — Participants will complete exposure therapy for up to 12 weeks, and coached exposure session will be approximately 50 minutes.

SUMMARY:
Exposure therapy is the most effective treatment available for obsessive compulsive disorder, yet up to 50% of patients do not recover because the mechanisms underlying successful response are poorly understood, leading to significant variability in how clinicians conduct exposure therapy. The main purpose of this study is to determine which target mechanisms are most critical to engage in real-world exposure sessions to produce good treatment outcomes. Adult participants (N = 400) with Obsessive Compulsive Disorder (OCD) receiving exposure therapy from two sites (McLean Hospital, San Diego State University) across the continuum of care (outpatient, partial hospital, residential) will complete baseline clinical and demographic measures as well as weekly symptom reports. The project will measure exposure mechanisms across three levels of analysis (self-report, observer-rated behavior, physiology) during each exposure session. Mechanisms assessed will include a broad range of variables based on both habituation and inhibitory learning models of exposure. Self-report and observer-rated mechanisms will be measured with the Exposure Feedback Form, created and piloted by the study team. Physiological mechanisms will include skin conductance response, heart rate, and heart rate variability measured with a wristwatch. The current study will determine (1) which exposure mechanisms lead to favorable clinical outcomes, and (2) what makes a good exposure for whom. Results of this study have the potential to improve personalized care for the many patients who do not remit following exposure therapy for OCD.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years old
* Seeking exposure treatment at McLean Hospital OCD Institute or San Diego State University
* Have a diagnosis of OCD
* Able to complete study measures and treatment procedures in English

Exclusion Criteria:

* Acute symptoms of psychosis
* Active suicidality (plan, means, intent and/or suicide attempt in past 3 months)
* Presence of co-occurring symptoms that warrant higher level of care (e.g., inpatient treatment)
* Presence of any medical, psychiatric, or developmental condition that would prevent patients from completing assessments or exposure exercises (e.g., non-verbal autism spectrum disorder)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (YBOCS) | Up to 12 weeks
  The YBOCS is a 10 self-report measure of OCD severity.

SECONDARY OUTCOMES:
Quality of Life Enjoyment & Satisfaction Questionnaire (QLES) | Up to 12 weeks
  The QLES is a 14-item self-report measure assesses the degree of enjoyment and satisfaction experienced in various daily functioning domains.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie M Kuckertz, PhD, Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - Center for Understanding and Treating Anxiety, San Diego, California
  - McLean OCDI, Belmont, Massachusetts